CLINICAL TRIAL: NCT03983733
Title: PREDICT 2: Personalized Responses to Dietary Composition Trial 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zoe Global Limited (Other)
Collaborators: Massachusetts General Hospital (Other); Stanford University (Other); King's College London (Other); Tufts University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PREDICT 2
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Diabetes; Heart Diseases; Diet Habit; Diet Modification; Microbial Colonization; Healthy; Obesity; Metabolism
Keywords: Gut microbiome; Personalised Nutrition; Metabolic health; Postprandial metabolism
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases; Feeding Behavior; Communicable Diseases; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention (Experimental): Dietary intervention using standardised test meals, on up to 8 days within the study period.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — To carry out an interventional dietary study using standardised meals to predict an individual's metabolic response to certain foods, using their gut microbiome, metabolic profile, and other measurable characteristics such as weight, sleep and exercise.

SUMMARY:
Foods in the human diet can affect the development of diseases over time, such as diabetes or heart disease. This is because the amount and types of foods in the diet eat can affect a person's weight, and because different foods are metabolised (processed) by the body in different ways.

Scientists have also found that the bacteria in the human gut (the gut microbiome) affect their metabolism, weight and health and that, together with a person's diet and metabolism, could be used to predict appetite and how meals affect the levels of sugar (glucose) and fats (lipids) found in blood after eating. If blood sugar and fat are too high too often for too long, there is a greater chance of developing diseases such as diabetes and cardiovascular disease.

The gut microbiome is different in different people. Only 10-20% of the types of bacteria found in the human gut are found in everyone. This might mean that the best diet to prevent disease needs matching to a person's gut microbiome and it might be possible to find personalised foods or diets that will help reduce the chance of developing chronic disease as well as metabolic syndrome.

The study investigators are recruiting volunteers aged 18-70 years to take part in a study that aims to answer the questions above. Participants will be asked to consume standardised meals on up to 8 days while wearing glucose monitors (Abbott Freestyle Libre) to measure their blood sugar levels. Participants will also be required to prick their fingers at regular intervals to collect small amounts of blood, and to record their appetite, food, physical activity and sleep using apps and wearable devices. They will be asked to collect a fecal and saliva sample before consuming the standardised meals, and to provide a fasted blood sample at the end of the study period.

DETAILED DESCRIPTION:
Choice of design: The study is a single arm mechanistic intervention study.

Study population: Participants will be recruited through online and offline advertisements, and through health professionals.

Screening Assessment: Prospective participants will be selected based on the defined inclusion and exclusion criteria by the study management team. Screening will be online and via phone. Prospective participants will be booked in to start their study period and will receive a study kit by post.

Study duration: Each participant will take part in the study for a period of up to 12 days.

Dietary intervention: The dietary intervention will be carried out on up to 8 days within the 12-day study period. On day one, participants will be asked to collect biological samples and fit wearable devices (glucose monitor and physical activity tracker). Over the following consecutive days, each participant will be instructed to eat up to 8 standardised meals for breakfast, which must be their first meal of the day. On up to 3 of the days the participants will also be asked to eat a standardised lunch. Participants are free to eat whatever they wish at all other times. The standardised meals will be provided to all participants by the study team via post. The foods included as part of these meals will be foods that are commonly consumed and can be made from products sold in US supermarkets. Participants will be reassured that the amount of food will be designed to ensure a stable body weight over the course of the study. Participants will be asked to consume the entire amount of food indicated for the standardised meals and to record any left-over food via a digital app for which training will be provided at the start of the study. Following completion of standardised meal days, participants are free to eat and drink whatever they wish and will be asked to track all meals, snacks and drinks on their digital app. Participants will also be advised not to change their physical activity patterns during the course of the study. The 12th day of the study involves a visit to a medical clinic where participants will provide a fasted blood sample.

Regular contact will be made with the participants via phone, their app and text messages for the period of the intervention to encourage compliance and answer any queries.

Anthropometry: The participant will be instructed to measure their weight, height, waist and hip circumference.

Dietary and Lifestyle: Participants will be asked to complete a baseline questionnaire online, as well as a diet history questionnaire with portion sizes about the month preceding their study period. They will be asked to record on a daily basis their dietary, activity, and psychological data (e.g. hunger) using a digital mobile phone app. Lifestyle information (such as sleep and exercise) will be monitored using digital wearable devices. Training in all apps and equipment will be given through written and online instructions and via communications with the study support staff.

Digital devices: Participants will be asked to record daily dietary and activity information using digital apps and lifestyle information will be monitored using digital wearable devices. The continuous glucose monitor (Freestyle Libre, CGM) provides continuous glucose profiles for up to 14 days. The CGM will be inserted on the back of the upper arm, one day before participants begin dietary intervention. This will measure subcutaneous interstitial fluid glucose concentrations every 5 minutes. The CGM will be removed at the end of the intervention period by the participant. A contact number will be made available to participants for any inquiries or if any problems arise. Data from the CGM will be downloaded, and glucose profiles will be evaluated on the basis of data collected.

Blood samples: The participant will collect postprandial blood on 2 days using finger-prick blood sampling. They will also provide a fasted blood sample after the study period to measure their baseline metabolomic profile.

Digital app: Participants will be asked to download an app designed specifically for this study, which provides diet & activity logging functionality similar to widely used existing apps such as MyFitnessPal.

Participants will be asked to record and monitor the following information via the digital app and wearable devices, on a daily basis:

* All food and drink they consume, with serving sizes and photos
* Sleep and physical activity patterns, including exercise
* Hunger and alertness ratings
* Psychological feeling of energy and mood
* Prescription and over-the-counter drug consumption

The app will be available in versions for both iOS and Android operating systems, and will support a wide range of mobile phone models as expected across the participant population. The app will synchronise remotely with backend database servers, over an encrypted and authenticated API, and will support offline operation for when patients wish to record an entry without network coverage. This continuous background synchronization means that it will not be necessary to explicitly download data from the phone at the end of the study.

Following the 2020 pandemic of COVID-19, participants are asked to use the COVID-19 Symptom Tracker app to record their physical health symptoms, or lack thereof, attributable to COVID-19, as well as demographic and other health information to track the spread of disease in real time, and to potentially reveal risk factors for infection and severe illness.

Subcohort: An opt-in follow-on study will be offered to participants to follow dietary guidance from the ZOE app based on their Predict 2 results. During the first 2 to 4 weeks, participants will be given dietary guidance to follow from the ZOE app. Thereafter, for a period of up to 12 months, participants will be asked to report on outcome measures at regular intervals (monthly). Outcome measures will be reported before, during and after the 2 to 4 week period and include weight, bristol stool, bowel habits, hunger, energy, alertness, stress, mood, activity, adherence to dietary advice, and app usage.

The data will be used to test the efficacy of the ZOE dietary advice in promoting weight loss and improvement of overall health, and may be stratified by age, sex, BMI, adherence and/or motivation to take part in the PREDICT 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-70 years of age (19 year age minimum in Alabama and Nebraska)
* Body mass index (BMI) between 16.5 and 49.9 kg/m2.
* Living in the continental USA.
* Able and willing to comply with the study protocol and provide informed consent.

Exclusion Criteria:

* Refuse or are unable to provide informed consent to participate in the study.
* Have ongoing, active inflammatory disease or condition e.g. Rheumatoid arthritis, systemic lupus erythematosus, polymyalgia and other connective tissue diseases.
* Have had cancer in the last two years, excluding skin cancer.
* Have been diagnosed with Inflammatory Bowel Disease (ulcerative colitis and Crohn's disease) or Celiac disease (gluten allergy), or any other long-term gastrointestinal disorder that would prevent the individual from safely eating normal US food. Irritable Bowel Syndrome is not an exclusion.
* Have had bariatric or other major gastrointestinal surgery.
* Have been medically advised that eating high-fat meals over a period of a few days might be dangerous.
* Currently suffer from severe anemia or jaundice.
* Have taken any of the following medications in the last three months:

immunosuppressants (including oral steroids) or antiretroviral therapies or antibiotics (excluding topical antibiotics). If diagnosed with non-alcoholic fatty liver disease, use of any steatogenic medications (amiodarone or methotrexate) or insulin in the last 3 months

* Have an uncontrolled intercurrent illness (e.g. hepatitis c, influenza)
* Are using proton pump inhibitors ("PPI"s such as omeprazole and pantoprazole), unless they are able to stop two weeks before the start of the study and abstain from use during the study.
* Have type 1 diabetes.
* Have type 2 diabetes and are taking insulin or sulfonyurea medications (such as Diamicron (Gliclazide), Diamicron MR (Gliclazide), Amaryl (Glimepiride), Daonil (Gilbenclamide or Glyburide), Gibenese (Glipizide), Minodiab (Glipizide), Tolbutamide (Tolbutamide)). For clarity, people with type 2 diabetes can participate if they take metformin or gliptins.
* Have type 2 diabetes and a fasting glucose level of >216mg/dL. These individuals wil be excluded whether or not they are on medication.
* Started antidepressant medication within the last 3 months, or are currently suffering from acute clinically diagnosed depression which is not well controlled.
* Have had a heart attack (myocardial infarction) or stroke in the last 6 months.
* Are pregnant or breastfeeding, have given birth in the last three months, or are planning to be pregnant in the next 3 months.
* Diagnosed with an eating disorder (e.g. anorexia nervosa or bulimia nervosa)
* Are vegan, or unwilling to consume foods that are part of the study.
* Do not have a mobile phone capable of running the Zoe study/results apps, or are unable to use their phone to operate the apps. As a consequence of this exclusion, all participants must be able to read and write in English, as the app is only available in English.
* Are unable to have continuous access to their smartphone or unable to wear the activity tracker on their arm for the duration of the study, e.g. because their work will not allow it.
* Have a known allergy to adhesives like that used to affix the continuous glucose monitor.
* Are unable or unwilling to visit a Quest center to provide fasting blood samples.
* Do not have access to wifi or unlimited mobile data to allow them to download the app for free and upload data during the study.
* Do not have a freezer to store study-related foods required for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Gut microbiome species richness | 1 Day
  Species count in fecal sample
Lipids | 3 days
  Measurement of blood lipids
Glucose | 11 days
  Measurement of blood glucose
Sleep | 10 days
  Record of sleep pattern using a wearable device (i.e. fitness watch)
Physical activity | 10 days
  Record of physical activity using a wearable device (i.e. fitness watch)
Hunger and appetite assessment | 10 days
  Record of hunger and appetite patterns using a digital app

SECONDARY OUTCOMES:
Glucose metabolism | 3 days
  C-peptide
Dietary assessment | 10 days
  Weighed food log
Anthropometry | 1 day
  Weight (kg)
Anthropometry | 1 day
  Height (cm)
Anthropometry | 1 day
  Hip and waist circumference (cm)
Metabolomics by NMR analysis | 1 day
  Lipoprotein concentration (mol/L), lipoprotein composition (mol/L), glycoprotein acetyl concentration (mol/L), ketone bodies concentration (mol/L)
Dietary assessment | 1 month
  Diet history and portion size questionnaire about the preceding month, using the Diet History Questionnaire 3 from National Cancer Institute.
Covid-19 symptom assessment | 6 months
  Self-reported demographic and physical health symptoms, or lack thereof, reported on a daily basis.

OTHER OUTCOMES:
Adherence (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on daily frequency of adherence (categorical)
Hunger (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on hunger levels (categorical)
Weight (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on weight (lbs)
Bristol Stool Category (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app Bristol Stool chart questoin (categorical)
Bowel Frequency (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on bowel frequency
Energy (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on energy levels (categorical)
Alertness (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on alertness (categorical)
Stress (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on stress (categorical)
Mood (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on mood (categorical)
Activity (in sub-cohort) | 12 months: Baseline, Weekly (0 to 4 weeks), monthly (5 to 24 weeks), 36 weeks, 52 weeks
  Self-reported in-app question on daily frequency of activity (categorical)
Dietary assessment | 12 months: 24 weeks, 52 weeks
  Diet history and portion size questionnaire about the preceding month, using the Diet History Questionnaire 3 from National Cancer Institute.
Gut microbiome species richness | 12 months: 24 weeks, 52 weeks
  Species count in fecal sample

CONTACTS AND LOCATIONS:
Overall Officials: Tim Spector, Pr., Principal Investigator — Zoe Global Limited
Locations (1):
- Zoe US Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No